CLINICAL TRIAL: NCT06686355
Title: Double-blind Randomized Parallel Contrast Clinical Study of Yiqilishui Formula on Sepsis Induced Myocardial Dysfunction
Brief Title: The Treatment of Sepsis Induced Myocardial Dysfunction With Yiqilishui Formula
Acronym: YQSIMD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Xiu Shengyao, Principal Investigator, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DongzhimenH
Record Dates: First submitted 2024-10-09; First posted 2024-11-13 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Sepsis Induced Myocardial Dysfunction
Keywords: sepsis; myocardial dysfunction; SIMD; Yiqilishui formula; Double-blind randomized; clinical study
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: Inclusion criteria:
  1. Patients hospitalized in the ICU of Beijing Tongzhou Traditional Chinese Medicine Hospital and the ICU of Dongzhimen Hospital of Beijing University of Traditional Chinese Medicine from January 2024 to December 2026.
  2. Meeting the diagnostic criteria for Qi deficiency and water overflow syndrome of septic cardiomyopathy.
  3. Age ≥50 and ≤80 years old;
  4. SOFA score: 2 to 12 points;
  5. Diagnosis of septic cardiomyopathy within 24 hours;
  6. Patient or family member has signed the informed consent form.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yiqilishui group (Experimental): Conventional Western medicine treatment + oral or nasogastric administration of Yiqilishui formula granules, twice daily;
  Interventions: Drug: Yiqilishui formula
- placebo group (Sham Comparator): Conventional Western medicine treatment + oral or nasal feeding of Yiqilishui formula placebo , twice daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Yiqilishui formula — Astragalus Root 30g, Angelica sinensis 30g, Honeysuckle Flower 30g, Capillary Artemisia Herb 15g, Giant Knotweed Rhizome 15g, Lepidium Seed 30g, Sichuan Lovage Rhizome 15g, Salvia Root 15g, Jujube Fruit 15g;
  Arms: Yiqilishui group
Other: Placebo — 5% Yiqilishui Granules + 95% Dextrin;
  Arms: placebo group

SUMMARY:
The goal of this clinical trial is to learn if Chinese medicine - Yiqilishui formula works to treat sepsis-induced myocardial dysfunction (SIMD). It will also learn about the safety of Yiqilishui formula. The main questions it aims to answer are:

* Compared with conventional western traetment alone, can supplementing conventional Western treatment with Yiqilishui formula better improve the heart function and reduce mortality of participants with SIMD?
* What medical problems do participants have when taking Yiqilishui formula? Researchers will compare Yiqilishui formula to a placebo (a look-alike substance that contains no drug) to see if Yiqilishui formula works to treat SIMD.

Participants will:

* Take Yiqilishui formula granules or placebo twice daily for 7 days, while receiving standard conventional Western treatment.
* Undergo blood drawing, electrocardiogram and transthoracic echocardiography at enrollment, on the 3rd day, the 7th day, and the 14th day after enrollment.

DETAILED DESCRIPTION:
Sepsis-induced myocardial dysfunction (SIMD) is characterized by high morbidity and mortality rates and remains a challenging issue in the field of critical care that has not yet been resolved. The main pathogenesis involves deficiency of Qi with water overflow and blood stasis and toxin blocking the channels. The use of a Qi-invigorating and diuretic formula has the effect of invigorating Qi, promoting diuresis, and detoxifying and unblocking the channels. This study employed a two-center prospective parallel randomized double-blind controlled trial, selecting a total of 80 SIMD subjects from the ICU of Tongzhou District Traditional Chinese Medicine Hospital and the ICU of Dongzhimen Hospital of Beijing University of Chinese Medicine, who met the inclusion and exclusion criteria. The subjects were randomly and evenly divided into a treatment group and a control group. Both groups received basic SIMD treatment, with the treatment group additionally receiving the oral or nasogastric administration of a granule preparation of Yiqilishui formula, and the control group receiving a placebo orally or nasogastrically. The intervention period was 7 days, with a follow-up period of 28 days. The primary efficacy indicators compared between the two groups were BNP and NT-proBNP, and the secondary efficacy indicators were echocardiography, myocardial injury markers, inflammatory markers, critical illness severity scores, ICU length of stay and costs, and 28-day survival rate. The study aimed to evaluate the clinical efficacy and safety of the Yiqilishui formula for SIMD.

ELIGIBILITY:
Inclusion Criteria

1. Patients hospitalized in the ICU of Tongzhou Traditional Chinese Medicine Hospital and Dongzhimen Hospital of Beijing University of Chinese Medicine between January 2024 and December 2026.
2. Patients diagnosed with SIMD and qi deficiency and water flooding syndrome.
3. Aged 50 to 80 years.
4. SOFA score: 2 to 12 points.
5. Diagnosis of SIMD within 24 hours.
6. Signed informed consent by the patient or their family.

Exclusion Criteria

1. Subjects diagnosed with acute coronary syndrome, old myocardial infarction, or those who have undergone coronary revascularization.
2. Subjects with heart failure caused by cardiomyopathies such as hypertrophic cardiomyopathy, dilated cardiomyopathy, myocardial amyloidosis, diabetic cardiomyopathy, or hypothyroid cardiomyopathy.
3. Subjects with heart failure caused by structural heart abnormalities, arrhythmias, pulmonary heart disease, or cardiorenal syndrome.
4. Subjects with severe primary diseases affecting survival, including uncontrolled, unresectable metastatic malignant tumors, hematologic diseases, and HIV.
5. Subjects with liver or kidney dysfunction, with an individual SOFA score of ≥3 for liver or kidney function.
6. Subjects who have used immunosuppressants continuously in the last 6 months or have undergone organ transplantation.
7. Subjects who have used corticosteroids (equivalent to methylprednisolone ≥20mg/day) continuously within 7 days prior to enrollment.
8. Subjects who have used Chinese herbal medicines or Chinese patent medicine replenishing qi, activating blood circulation and facilitating diuresis within 14 days prior to enrollment.
9. Subjects deemed unable to take decoctions by clinicians.
10. Pregnant or breastfeeding women.
11. Subjects with a body mass index (BMI) <18.5 or >30.
12. Subjects who have participated in other clinical trials within the last 30 days.
13. Subjects deemed unable to complete or unsuitable for this study by the researchers (e.g., expected death within 48 hours or refusal of active treatment).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
BNP（B-type natriuretic peptide） decline rate | At enrollment, on the 3rd day, the 7th day, and the 14th day
  Blood samples were taken from the median cubital vein of the subjects at enrollment, on the 3rd day, the 7th day, and the 14th day to measure the BNP levels in the subjects' venous blood, calculate the patient's BNP decline rate, assess the severity of heart failure in the subjects, and predict their prognosis.

SECONDARY OUTCOMES:
The levels of cTnI | At enrollment, on the 3rd day, the 7th day, and the 14th day
  Cardiac injury markers-Blood samples from the median cubital vein of the subjects were taken at enrollment, on the 3rd day, the 7th day, and the 14th day to detect the levels of cardiac troponin I (cTnI)
The levels of CK-MB | At enrollment, on the 3rd day, the 7th day, and the 14th day
  Cardiac injury markers-Blood samples from the median cubital vein of the subjects were taken at enrollment, on the 3rd day, the 7th day, and the 14th day to detect the levels of creatine kinase MB isoenzyme
Concentration of H-FABP | At enrollment, on the 3rd day, the 7th day, and the 14th day
  Cardiac injury markers-Blood samples from the median cubital vein of the subjects were taken at enrollment, on the 3rd day, the 7th day, and the 14th day to detect the levels of heart-type fatty acid-binding protein
Tei index | At enrollment, on the 3rd day, the 7th day, and the 14th day
  At the time of subject enrollment, on the 3rd day, 7th day, and 14th day, Tei index were measured using transthoracic echocardiography to evaluate the subjects' cardiac function and structure.
MEE | At enrollment, on the 3rd day, the 7th day, and the 14th day
  At the time of subject enrollment, on the 3rd day, 7th day, and 14th day, myocardial energy expenditure
LVMI | At enrollment, on the 3rd day, the 7th day, and the 14th day
  At the time of subject enrollment, on the 3rd day, 7th day, and 14th day, left ventricular mass index (LVMI) were measured using transthoracic echocardiography to evaluate the subjects' cardiac function and structure.
The levels of WBC | At enrollment, on the 3rd day, the 7th day, and the 14th day
  Blood is drawn from the median cubital vein of the subjects at enrollment, on the 3rd day, the 7th day, and the 14th day. The levels of white blood cells (WBC) in the subjects' venous blood is detected.
The percentage of NE% | At enrollment, on the 3rd day, the 7th day, and the 14th day
  Blood is drawn from the median cubital vein of the subjects at enrollment, on the 3rd day, the 7th day, and the 14th day. The percentage of neutrophils (NE%) in the subjects' venous blood is detected.
The levels of CRP | At enrollment, on the 3rd day, the 7th day, and the 14th day
  Blood is drawn from the median cubital vein of the subjects at enrollment, on the 3rd day, the 7th day, and the 14th day. The levels of C-reactive protein (CRP) in the subjects' venous blood is detected.
The levels of PCT | At enrollment, on the 3rd day, the 7th day, and the 14th day
  Blood is drawn from the median cubital vein of the subjects at enrollment, on the 3rd day, the 7th day, and the 14th day. The levels of procalcitonin (PCT) in the subjects' venous blood is detected.
Concentration of IL-6 | At enrollment, on the 3rd day, the 7th day, and the 14th day
  The supernatant serum is obtained by centrifugation, and the levels of interleukin-6 (IL-6) is measured by ELISA.
Concentration of TNF-α | At enrollment, on the 3rd day, the 7th day, and the 14th day
  The supernatant serum is obtained by centrifugation, and the levels of tumor necrosis factor-α (TNF-α) is measured by ELISA.
Concentration of ROS | At enrollment, on the 3rd day, the 7th day, and the 14th day
  The supernatant serum is obtained by centrifugation, and reactive oxygen species (ROS)is measured by ELISA.
Concentration of ATP | At enrollment, on the 3rd day, the 7th day, and the 14th day
  The supernatant serum is obtained by centrifugation, and the levels of ATP content in the subjects' serum is measured by ELISA.
Platelet aggregation rate | At enrollment, on the 3rd day, the 7th day, and the 14th day
  At enrollment, D3, D7, and D14, venous blood from patients is collected, platelet-rich plasma is prepared using differential centrifugation, and the platelet aggregation rate is determined by optical turbidimetry.
SOFA score | At enrollment, the 7th day, and the 14th day
  Sequential Organ Failure Assessment (SOFA score) is performed at the time of enrollment, on the 7th day, and on the 14th day. The SOFA score includes six systems: respiratory, circulation, liver, coagulation, kidney and central nervous system. Each system is scored according to different variables, with a score of 0 to 4 points, and a total score of 0 to 24 points. The higher the score, the worse the outcome.
Apache II score | At enrollment, the 7th day, and the 14th day
  Acute Physiology and Chronic Health Evaluation (Apache II score) is performed at the time of enrollment, on the 7th day, and on the 14th day. The Apache II score is scored from 0 to 71, and the higher the score, the worse the outcome.
ICU length of stay; | From the date the participant is transferred to the ICU to the date he or she is finally transferred out of the ICU, assessed up to 100 weeks.
  ICU length of stay，up to 100 weeks.
Outcome indicator | 28th day
  28-day mortality rate

OTHER OUTCOMES:
The level of body temperature | Daily from enrollment to the 7th day.
  During the intervention period, record the patient's underarm temperature measurement daily.
Breathing rate | Daily from enrollment to the 7th day.
  During the intervention period, record the patient's breathing rate measurement daily.
Heart rate | Daily from enrollment to the 7th day.
  During the intervention period, record the patient's heart rate measurement daily.
The levels of blood pressure | Daily from enrollment to the 7th day.
  During the intervention period, record the patient's blood pressure measurement daily.
The levels of ALT | At enrollment and on the 7th day.
  Before and after intervention period, record the patient's the levels of ALT.
The levels of AST | At enrollment and on the 7th day.
  Before and after intervention period, record the patient's the levels of AST.
The levels of BUN | At enrollment and on the 7th day.
  Before and after intervention period, record the patient's the levels of BUN.
The levels of Cr | At enrollment and on the 7th day.
  Before and after intervention period, record the patient's the levels of Cr.
The levels of PT | At enrollment and on the 7th day.
  Before and after intervention period, record the patient's the levels of Prothrombin Time(PT).
The levels of APTT | At enrollment and on the 7th day.
  Before and after intervention period, record the patient's the levels of Activated Partial Thromboplastin Time(APTT).
The levels of INR | At enrollment and on the 7th day.
  Before and after intervention period, record the patient's the levels of international normalized ratio(INR).
The levels of TT | At enrollment and on the 7th day.
  Before and after intervention period, record the patient's the levels of Thrombin Time(TT).
The levels of D-D | At enrollment and on the 7th day.
  Before and after intervention period, record the patient's the levels of D-dimer(D-D).
The levels of FDP | At enrollment and on the 7th day.
  Before and after intervention period, record the patient's the levels of Fibrin degradation products(FDP).
Unexpected adverse reactions | From enrollment to the 7th day, unexpected adverse reactions should be recorded at any time during the intervention period.
  Unexpected adverse reactions occurred during the intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongzhimen Hospital Affiliated to Beijing University of Chinese Medicine, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes